CLINICAL TRIAL: NCT00559234
Title: Evaluation and Treatment Protocol for Potential Research Participants With Inherited Ophthalmic Diseases
Brief Title: Potential Research Participants for Future Studies of Inherited Eye Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080017; 08-EI-0017
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-03

CONDITIONS: Cataract; Glaucoma; Retinitis Pigmentosa; Macular Degeneration; Strabismus
Keywords: Optic Nerve; Retina; Cornea; Lens; Ocular Genetic Diseases; Inherited Eye Disease; Genetic Eye Disease
MeSH Terms: conditions — Cataract; Glaucoma; Retinitis Pigmentosa; Macular Degeneration; Strabismus; Corneal Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will evaluate potential candidates for future clinical research studies related to diagnosed or undiagnosed genetic eye disorders or diseases. It will not test any new treatments, but it may arrange for standard treatments for existing eye disorders. The purpose of the study is to train eye doctors and medical researchers at the National Institutes of Health in appropriate methods and procedures for treating patients with genetic eye diseases, and to expand the pool of possible participants for future research studies and trials on eye health.

Volunteers for this study may be adults and minor children who have been diagnosed with or are at risk for having a genetic eye disease. Candidates may not have any other medical conditions that would interfere with the researchers' ability to perform the examinations and procedures required for this study.

Participants will give a complete medical and family history and undergo a series of tests and procedures as part of this research study. The procedures include a full eye examination and vision testing, electrooculography and an electroretinogram to examine the function of the retina, and flourescein angiography to provide information on the flow of blood in the participant's eyes. Participants will provide research material for further studies by giving a blood sample to be held for genetic testing and analysis, and adult participants will also undergo a skin biopsy to provide cell tissue for additional research material. At each clinic visit, participants will receive treatment for their genetic eye disease as needed, including medications or surgical procedures. Participants may remain a part of this study for up to three years.

DETAILED DESCRIPTION:
The National Eye Institute is conducting a study to evaluate participants with either diagnosed or undiagnosed genetic conditions who may be eligible and wish to participate in other NEI clinical research studies. The primary purpose of this evaluation and treatment protocol is to provide a resource of patients for specific new research protocols and for staff and fellowship training. A secondary purpose is to provide long-term follow-up and treatment for a variety of genetic eye diseases so that the genetic specialists at NEI will be better able to identify research hypotheses for these diseases, which may lead to ideas for future protocols. Finally, the ability to provide long-term follow-up and care will also facilitate referral efforts for new NEI protocols. As a by-product of this research activity, the participants will help the investigators to maintain their clinical skills.

ELIGIBILITY:
* INCLUSION CRITERIA

Subjects will be able to enroll if they:

* Have either a diagnosed or undiagnosed genetic eye disease.
* Have the ability to understand and sign an informed consent or have a parent/legal guardian who is able to do so for them.

EXCLUSION CRITERIA

Subjects will not be eligible if they:

* Are unwilling or unable to be followed and treated at the NEI Clinical Center.
* Have any systemic diseases that compromise the ability to provide adequate ophthalmologic examination or treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2007-11-09; Study Completion 2008-10-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] MacDonald IM, Mah DY. Summary of heritable ocular disorders and selected systemic conditions with eye findings. Ophthalmic Genet. 2000 Mar;21(1):29-49. PMID 10779848
- [Background] MacDonald IM, Haney PM, Musarella MA. Summary of ocular genetic disorders and inherited systemic conditions with eye findings. Ophthalmic Genet. 1998 Mar;19(1):1-17. doi: 10.1076/opge.19.1.1.2181. PMID 9587925